CLINICAL TRIAL: NCT05614258
Title: A First-in-Human (FIH), Open-Label, Phase 1 Study of ADG206, a CD137 Agonist Antibody, in Subjects With Advanced/Metastatic Solid Tumors
Brief Title: Study of ADG206 in Subjects With Advanced/Metastatic Solid Tumors
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Adagene Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ADG206-1001
Record Dates: First submitted 2022-10-27; First posted 2022-11-14 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Advanced/Metastatic Solid Tumors

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ADG206 dose escalation (Experimental)
  Interventions: Drug: ADG206

INTERVENTIONS:
Drug: ADG206 — All participants in this study will receive the study drug ADG206 in one of the designed dosage level. ADG206 will be administered by intravenous infusion over 60-90 minutes on Day 1 of each treatment cycle until disease progression, intolerable toxicities or withdrawal of consent, or up to 2 years.

SUMMARY:
ADG206 is an activatable prodrug form of a fully human monoclonal antibody (mAb) of the immunoglobulin G1 (IgG1) subclass that specifically targets cluster of differentiation 137 (CD137) (also known as 4-1BB) as a co-stimulatory receptor agonist for the treatment of advanced malignancies.

DETAILED DESCRIPTION:
This is a FIH, Phase 1, open-label, multicenter, sequential dose escalation study to evaluate the safety, tolerability, Pharmacokinetics (PK), and preliminary efficacy of ADG206 in subjects with advanced/metastatic malignancies.

Primary Objective of the study: To assess safety and tolerability at increasing dose levels of ADG206 in subjects with advanced/metastatic solid tumors who have exhausted their treatment alternatives.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status ≤1.
* Subjects with advanced or metastatic solid tumors (except thymic tumors), which have progressed after all standard therapies, or no further standard therapies exists.
* At least 1 measurable lesion per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1).
* Adequate organ function.
* Woman of childbearing potential must agree to use 2 methods of acceptable contraception from screening until 6 months after the last dose of study drug.
* Male subjects who are sexually active with a female partner of childbearing potential must agree to use a barrier contraception.

Exclusion Criteria:

* Subjects within washout period of other anti-tumor therapies. .
* History of prior malignancy other than the cancer under treatment in the study.
* Major trauma or major surgery within 4 weeks before the first dose of study drug.
* Serious nonhealing wound, ulcer, or bone fracture.
* History of significant immune-mediated AE.
* Central nervous system (CNS) disease involvement.
* Any evidence of underlying severe liver dysfunction.
* Prior organ allograft transplantations or allogeneic bone marrow, cord blood or peripheral blood stem cell transplantation.
* Clinically significant cardiac disease with insufficient cardiac function.
* Evidence of active uncontrolled viral, bacterial, or systemic fungal infection.
* Known positive test result for human immunodeficiency virus (HIV) or acquired immune deficiency syndrome (AIDS).
* Infection of hepatitis B virus (HBV), or hepatitis C virus (HCV) (unless the disease is clinically controlled) .
* History or risk of autoimmune disease.
* Subjects with active severe lung infection or with a history of interstitial lung diseases, noninfectious pneumonitis, active pulmonary tuberculosis, or evidence of active pneumonitis. Clinically significant and unmanageable ascites defined as requiring constant therapeutic paracentesis.
* Any serious underlying issue that would limit compliance with study requirements, impair the ability of the subject to understand informed consent.
* Known hypersensitivity, allergies, or intolerance to immunoglobulins or to any excipient contained in ADG206.
* Pregnant, lactating, or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2023-02-13 (Actual); Primary Completion 2025-06-25 (Actual); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants experiencing dose-limiting toxicities escalating dose levels | At the end of Cycle 1 (each cycle is 21 days)
Number of participants with adverse events (AE) | At the end of 90 days post last dose (each cycle is 21 days)
Maximum administered dose (MAD) of ADG206 | At the end of the last dose (each cycle is 21 days)
Maximum tolerated dose (MTD) of ADG 206 | At the end of the last dose (each cycle is 21 days)
Recommended Phase 2 dose (RP2D) of ADG206 | At the end of the last dose (each cycle is 21 days)

SECONDARY OUTCOMES:
The area under the curve (AUC) of plasma concentration of drug | At the end of the last dose (each cycle is 21 days)
Immunogenicity endpoints include antidrug antibodies (ADAs) | At the end of the last dose (each cycle is 21 days)
Maximum concentration (Cmax) | At the end of the last dose (each cycle is 21 days)
Time to maximum plasma concentration (Tmax) | At the end of the last dose (each cycle is 21 days)
Lowest plasma concentration (C[trough]) | At the end of the last dose (each cycle is 21 days)

CONTACTS AND LOCATIONS:
Locations (2):
- Australia (2):
  - Ashford Cancer Centre Research, Kurralta Park, South Australia
  - Monash Health, Clayton, Victoria

IPD SHARING:
Plan to Share IPD: No